CLINICAL TRIAL: NCT06582134
Title: Effectiveness of Brief Mindfulness-Based Interventions (BMBI) for Painful Temporomandibular Disorders (TMD) Among University Students
Brief Title: Effectiveness of Brief Mindfulness-Based Interventions for Painful Temporomandibular Disorders Among University Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Chan Siew Wui, Dr., University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DF OS2309/0063 (P)
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Temporomandibular Disorders; Chronic Pain
Keywords: Brief mindfulness-based intervention; Temporomandibular disorders; University students
MeSH Terms: conditions — Temporomandibular Joint Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Sham Comparator): Three 10-minute audio recordings (1, 2, 3) in MPEG-1 Audio Layer 3 (MP3) format consisting of relaxing music that mimic BMBI in duration but do not contain instructions specific to mindfulness training.
  Interventions: Behavioral: Sham BMBI
- Brief Mindfulness-Based Intervention (Experimental): Three 10-minute audio recordings (A,B,C) for BMBI in MPEG-1 Audio Layer 3 (MP3) format that contain mindfulness training based on the breathing concept in a background of relaxing music.
  Interventions: Behavioral: BMBI

INTERVENTIONS:
Behavioral: Sham BMBI — Participants are requested to listen to the recordings 3 times a week, for 3 months (in a standardized sequence e.g., 1-2-3 and repeat) on Mondays-Wednesdays-Fridays. They are instructed to listen right before they sleep and encouraged to use them whenever they feel stressed or in pain.
  Arms: Control
Behavioral: BMBI — Participants are requested to listen to the recordings 3 times a week, for 3 months (in a standardized sequence e.g. A-B-C and repeat) on Mondays-Wednesdays-Fridays. They are instructed to listen right before they sleep and encouraged to use them whenever they feel stressed or in pain.
  Arms: Brief Mindfulness-Based Intervention

SUMMARY:
The goal of this clinical trial is to learn if brief mindfulness-based intervention (BMBI) is beneficial to participants suffering from painful temporomandibular disorders (TMD). The objectives of the research are:

1. To compare physical functioning (pain intensity and jaw function) in UM students with chronic pain-related TMD before and after receiving BMBI
2. To compare psychological distress and mindfulness state in UM students with chronic pain-related TMD before and after receiving BMBI
3. To compare the quality of life of UM students with chronic pain-related TMD before and after receiving BMBI
4. To compare the changes in physical functioning, psychological distress, mindfulness state and quality of life between UM students in the intervention (BMBI) and the control groups.

Participants will:

Listen to the audio recordings 3 times a week, for 3 months when they are about to sleep.

Make 4 visits to the clinic: Baseline, 2 weeks, 1 month and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* Students attending Universiti Malaya
* Able to read and understand English.
* Willing and able to give informed consent.
* Score 3 and above on the TMD-PS, for at least 3 months.

Exclusion Criteria:

* Hearing impairment.
* Currently on psychiatric follow up and/or taking psychotropic prescriptions (antidepressants, anti-anxiety medications, stimulants, antipsychotics, and mood stabilizers).
* Experience with activities similar to the intervention such as meditation, yoga or tai chi.
* Currently practicing some form of mindfulness meditation.
* History of orofacial trauma, craniofacial pathology, and previous orofacial surgeries (including orthognathic and TMJ)
* Systemic rheumatic, neurologic/neuropathic, endocrine (e.g., diabetes mellitus) or immune / autoimmune diseases or widespread pain or being treated with immunosuppressant drugs
* Non-TMD orofacial pain disorders
* Radiation treatment to head and neck.
* Use of narcotic pain medication, muscle relaxants or steroid therapy unless discontinued 1 week before enrolment to study
* Use of nonsteroidal anti-inflammatory medications unless the medication(s) were discontinued for 3 days prior to enrolment (use of acetaminophen is allowed as a rescue drug)
* Currently on antibiotics or taken antibiotics within the last 2 weeks prior to start of study
* Currently pregnant or lactating women

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Degree of Pain Intensity | Change from Baseline at 2 weeks, 1 month and 3 Months
  * Graded Chronic Pain Scale Version 2.0 (GCPS v2)
  * 3 items for Characteristic Pain Intensity (CPI), 4 items for Interference Score and 1 item for Disability points for number of days with interference
  * CPI and Interference Scores are derived from computed mean of items, multiply by 10
  * Disability points for number of days with interference is determined from assigned points in a designated table
  * Total Disability Points = points for Disability Days + points for Interference Score
  * CPI and Disability Points will determine chronic pain grade (1=none; I=low intensity pain, without disability; II=high intensity pain, without disability; III- moderately limiting; IV=severely limiting)
Degree of Limitation of Jaw Function | Change from Baseline at 2 weeks, 1 month and 3 Months
  * Jaw Function Limitation Scale (JFLS-8) questionnaire
  * 8-item global scale for overall functional limitation of the masticatory system
  * Each item is rated on a numerical rating scale of 0 to 10 (0 indicates no limitation; 10 indicates severe limitation)
  * Mean of available items will determine degree of limitation
Level of Psychological distress | Change from Baseline at 2 weeks, 1 month and 3 Months
  * Psychological Distress (PHQ-4) questionnaire
  * 4 items, each with scores ranging from 0 (not at all) to 3 (nearly every day)
  * total score ≤2 indicates none-to-minimal levels of depression or anxiety, 3 to 5 indicates mild levels, 6 to 8 indicates moderate levels and ≥9 indicates severe levels
Extent of Impact on Oral-health Related Quality of Life | Change from Baseline at 2 weeks, 1 month and 3 Months
  * Oral Health Impact Profile-TMD (OHIP-TMD-22)
  * 22 items tool assessing oral health-related quality of life specific to TMD
  * Responses are scored from 0-4: never (0), hardly ever (1), occasionally (2), often(3), and very often (4)
  * Sum of scores ranges from 0 to 88 points, with higher scores indicating poorer quality of life

SECONDARY OUTCOMES:
Mindfulness state | Change from Baseline at 2 weeks, 1 month and 3 Months
  * Five Facet Mindfulness questionnaire (FFMQ-15)
  * 15 items assessing 5 facets (Observing, Describing, Acting with Awareness, Non-Judging of inner experience, Non-Reactivity to inner experience), with 3 items per facet
  * Results consist of a total average score and five subscales. Average scores are calculated by summing the responses and dividing by the number of items and indicate the average level of agreement with each subscale (1 = rarely true, 5 = always true). Higher scores indicate greater mindfulness.

OTHER OUTCOMES:
Width of Mouth Opening | Change from Baseline at 2 weeks, 1 month and 3 Months
  - Measurement of interincisal distance on reference teeth during maximum mouth opening without pain, with pain and with assistance
Number of Palpation Sites With Pain | Change from Baseline at 2 weeks, 1 month and 3 Months
  * number of palpation sites (temporomandibular joint and muscles) that is painful
  * muscles palpation: temporalis, masseter, posterior mandibular region, submandibular region, lateral pterygoid area, temporalis tendon)

CONTACTS AND LOCATIONS:
Overall Officials: Kathreena Kadir, MClinDent (OMFS)(Mal), Study Chair — Faculty of Dentistry, Universiti Malaya
Locations (1):
- Oral Medicine Clinic, Faculty of Dentisty, Universiti Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang D, Lee EKP, Mak ECW, Ho CY, Wong SYS. Mindfulness-based interventions: an overall review. Br Med Bull. 2021 Jun 10;138(1):41-57. doi: 10.1093/bmb/ldab005. PMID 33884400
- [Background] McClintock AS, McCarrick SM, Garland EL, Zeidan F, Zgierska AE. Brief Mindfulness-Based Interventions for Acute and Chronic Pain: A Systematic Review. J Altern Complement Med. 2019 Mar;25(3):265-278. doi: 10.1089/acm.2018.0351. Epub 2018 Dec 5. PMID 30523705
- [Background] Schumer MC, Lindsay EK, Creswell JD. Brief mindfulness training for negative affectivity: A systematic review and meta-analysis. J Consult Clin Psychol. 2018 Jul;86(7):569-583. doi: 10.1037/ccp0000324. PMID 29939051
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Yule PL, Durham J, Playford H, Moufti MA, Steele J, Steen N, Wassell RW, Ohrbach R. OHIP-TMDs: a patient-reported outcome measure for temporomandibular disorders. Community Dent Oral Epidemiol. 2015 Oct;43(5):461-70. doi: 10.1111/cdoe.12171. Epub 2015 Jun 4. PMID 26040190
- [Background] Baer RA, Carmody J, Hunsinger M. Weekly change in mindfulness and perceived stress in a mindfulness-based stress reduction program. J Clin Psychol. 2012 Jul;68(7):755-65. doi: 10.1002/jclp.21865. Epub 2012 May 23. PMID 22623334
- See also: Diagnostic Criteria for Temporomandibular Disorders: Scoring Manual for Self-Report Instruments. — https://ubwp.buffalo.edu/rdc-tmdinternational/tmd-assessmentdiagnosis/dc-tmd/